CLINICAL TRIAL: NCT01290939
Title: Phase III Trial Exploring the Combination of Bevacizumab and Lomustine in Patients With First Recurrence of a Glioblastoma
Brief Title: Bevacizumab and Lomustine for Recurrent GBM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-26101; EORTC-26101 (Other: EORTC); EU-21103; 2010-023218-30 (EudraCT Number); MO22968 (Other: F. Hoffmann-La Roche Ltd)
Record Dates: First submitted 2011-02-04; First posted 2011-02-07 (Estimated); Last update posted 2021-02-15 (Actual); Status verified 2021-02

CONDITIONS: Glioblastoma Multiforme; Cognition Disorders; Disability Evaluation
Keywords: adult glioblastoma; recurrent adult brain tumor; Cognition Disorders; functional defects
MeSH Terms: conditions — Glioblastoma; Cognition Disorders; Brain Neoplasms | interventions — Bevacizumab; Lomustine; DNA Methylation; Mental Status and Dementia Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): Lomustine 90 mg/m² every 6 weeks (cap. 160 mg) + bevacizumab 10 mg/kg every 2 weeks (at further progression treatment will be according to investigators discretion). In the absence of hematological toxicity > grade 1 during the first cycle the dose of lomustine can be escalated to 110 mg/m² (cap 200 mg) in their second cycle.
  Interventions: Biological: bevacizumab; Drug: lomustine; Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: cognitive assessment; Procedure: quality-of-life assessment
- Arm 2 (Active Comparator): Lomustine single agent 110 mg/m² every 6 weeks (cap. 200 mg) (at further progression treatment will be according to investigators discretion).
  Interventions: Drug: lomustine; Genetic: DNA methylation analysis; Other: laboratory biomarker analysis; Procedure: cognitive assessment; Procedure: quality-of-life assessment

INTERVENTIONS:
Biological: bevacizumab
  Arms: Arm 1
Drug: lomustine
Genetic: DNA methylation analysis
Other: laboratory biomarker analysis
Procedure: cognitive assessment
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Drugs used in chemotherapy, such as lomustine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. It is not yet known which regimen of bevacizumab given together with lomustine is most effective in treating patients with glioblastoma multiforme in first recurrence.

PURPOSE: The primary objective of this study is to investigate whether the addition of bevacizumab to lomustine improves overall survival (OS) in patients with recurrent glioblastoma compared to treatment with lomustine alone.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the therapeutic role of bevacizumab as well as the most favorable approach to treatment optimization for sequencing the combination of bevacizumab and lomustine in patients with glioblastoma multiforme in first recurrence.

OUTLINE: This is a multicenter study. Patients are stratified according to institution, WHO performance status (0 vs > 0), steroid administration (yes vs no), and largest diameter of tumor (≤ 40 mm vs > 40 mm). Patients are randomized at 2:1 ratio to 1 of 2 treatment arms.

* Arm 1: Lomustine 90 mg/m² every 6 weeks (cap. 160 mg) + bevacizumab 10 mg/kg every 2 weeks (at further progression treatment will be according to investigators discretion). In the absence of hematological toxicity > grade 1 during the first cycle the dose of lomustine can be escalated to 110 mg/m² (cap 200 mg) in their second cycle.
* Arm 2 (control arm): Lomustine single agent 110 mg/m² every 6 weeks (cap. 200 mg) (at further progression treatment will be according to investigators discretion).

One cycle will be defined arbitrarily (due to the lomustine sequencing) as 6 weeks for all arms. Day 1 of a cycle will be the first day when medication is taken.

Previously collected blood and tumor tissue samples are analyzed for MGMT methylation status, isocitrate dehydrogenase 1, and biomarkers of the VEGF pathway.

Patients and their caregivers/relatives complete quality-of-life questionnaires (EORTC QLQ-C30 and EORTC-BN20) at baseline, at 12 weeks, and then every 12 weeks after completion of study therapy. Patients also undergo neurocognitive assessment at baseline, at 12 weeks, and then every 12 weeks after completion of study therapy.

After completion of study treatment, patients are followed every 12 weeks.

ELIGIBILITY:
Histologically confirmed de novo glioblastoma (primary) with unequivocal first progression after RT concurrent/adjuvant chemotherapy at least 3 months off the concomitant part of the chemoradiotherapy

* Availability of biological material (tumor) for central review processes and translational research projects (tumor and blood)
* No more than one line of chemotherapy (concurrent and adjuvant temozolomide based chemotherapy including in combination with another investigational agent is considered one line of chemotherapy). Chemotherapy must have been completed at least 4 weeks prior to randomization if prior temozolomide
* No current or recent (within 4 weeks before randomization) treatment with another investigational drug
* No prior treatment with bevacizumab or other VEGF inhibitors or VEGF-Receptor signaling inhibitors
* No prior treatment with nitrosoureas
* Patient may have been operated for recurrence. If operated:
* residual and measurable disease after surgery is not required but surgery must have confirmed the recurrence
* a post-surgery MRI should be available within 48 hours following surgery
* Surgery completed at least 2 weeks before randomization and patients should have fully recovered
* Craniotomy or intracranial biopsy site must be adequately healed free of drainage or cellulitis, and the underlying cranioplasty must appear intact at the time of randomization.
* Study treatment should be initiated > 28 days following the last surgical procedure (including biopsy, surgical resection, wound revision, or any other major surgery involving entry into a body cavity)
* For non operated patients recurrent disease must be at least one bi-dimensionally measurable contrast-enhancing lesion with clearly defined margins by MRI scan, with minimal diameters of 10 mm, visible on 2 or more axial slices 5 mm apart, based on MRI scan done within two weeks prior to randomization
* Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
* Patients who require anti-convulsant therapy must be taking non-enzyme inducing antiepileptic drugs (non-EIAED). Patients previously on EIAED must be switched to non-EIAED at least 2 weeks prior to randomization
* No non tumor related surgery or other invasive procedures (major surgical procedure, open biopsy or significant traumatic injury) within 4 weeks prior to randomization, or anticipation of the need for major surgery during the course of the study treatment.
* No core biopsy or other minor surgical procedure within 7 days prior to randomization. Placement of a central vascular access device (CVAD) if performed at least 2 days prior to study treatment administration is allowed
* No radiotherapy within the three months prior to the diagnosis of progression
* No radiotherapy with a dose over 65 Gy, stereotactic radiosurgery or brachytherapy unless the recurrence is histologically proven No previous other malignancies, except for any previous malignancy which was treated with curative intent more than 5 years prior to randomization, and except for adequately controlled limited basal cell carcinoma of the skin, squamous carcinoma of the skin or carcinoma in situ of the cervix
* Absence of any cardiovascular disorder, including but not limited to:
* No history of myocardial infarction, unstable angina within 6 months prior to randomization
* No "New York Heart Association" (NYHA) Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication.
* No significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
* No prior history of hypertensive crisis or hypertensive encephalopathy
* No inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 m Hg)
* Absence of any thrombotic or hemorrhagic event, including but not limited to:
* No evidence of recent hemorrhage on MRI of the brain. However, patients with clinically asymptomatic presence of hemosiderin depositions, resolving hemorrhagic changes related to surgery, and presence of punctate hemorrhage in the tumor are permitted entry into the study
* No history or evidence of inherited bleeding diathesis or coagulopathy with the risk of bleeding.
* No arterial or venous thrombosis ≤ 6 months prior to randomization
* No history of stroke or TIAs within 6 months prior to randomization
* No history of pulmonary haemorrhage/haemoptysis ≥ grade 2 according to the NCI-CTCAE version 4.0 criteria within 1 month prior to randomization
* Absence of current or recent (within 10 days of first dose of bevacizumab) use of aspirin (> 325 mg/day) or other NSAID with anti-platelet activity or treatment with dipyramidole, ticlopidine, clopidogrel or cilostaz.
* International normalized ratio (INR) > 1.5 ULN and activated partial thromboplastin time (aPTT) > 1.5 × the ULN. Use of full-dose anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard in the institution) and the patient has been on a stable dose of anticoagulants for at least two weeks before randomization. As per ASCO guidelines, LMWH should be the preferred approach.
* Absence of known hypersensitivity:
* to any part of the bevacizumab or lomustine formulations.
* to Chinese hamster ovary cell products or other recombinant human or humanized antibody.
* No underlying or previous conditions that could interfere with treatment, including but not limited to:
* No history of intracranial abscess within 6 months prior to randomization
* No clinically serious (as judged by the investigator) non-healing wounds, active skin ulcers or incompletely healed bone fracture.
* No history of active gastroduodenal ulcer(s).
* No history of abdominal fistula as well as non-GI fistula, gastrointestinal perforation or intra-abdominal abscess within 6 months prior to inclusion.
* No evidence of active infection requiring hospitalization or antibiotics, within 2 weeks prior to randomization.
* No other diseases, interfering with follow up.
* Normal hematological functions: neutrophils ≥ 1.5 x 109 cells/l, platelets ≥ 100 x 109 cells/l and Hb ≥ 6.2 mmol/l (9.9 g/dl).
* Normal liver function: bilirubin < 1.5 x upper limit of the normal range (ULN), alkaline phosphatase and transaminases (ASAT) < 2.5 x ULN.
* Normal renal function: calculated (Cockcroft-Gault) or measured creatinine clearance > 30 mL/min; Urine dipstick for proteinuria < 2+. Patients with ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo 24 hours urine collection and must demonstrate ≤ 1 g of protein/24 hr.
* Age ≥ 18 years
* WHO Performance status 0 - 2
* Absence of pregnancy. Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and 6 months beyond stop of treatment in such a manner that the risk of pregnancy is minimized. In general, the decision for appropriate methods to prevent pregnancy should be determined by discussions between the investigator and the study subject. WOCBP include any female who has experienced menarche and who has not undergone successful surgical sterilization (hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or is not postmenopausal. Females should not be breast feeding.
* Post menopause is defined as: amenorrhea ≥ 12 consecutive months without another cause or for women with irregular menstrual periods and on hormone replacement therapy (HRT), a documented serum follicle stimulating hormone (FSH) level > 35 mIU/mL
* Women who are using oral contraceptives, other hormonal contraceptives (vaginal products, skin patches, or implanted or injectable products), or mechanical products such as an intrauterine device or barrier methods (diaphragm, condoms, spermicide) to prevent pregnancy, or are practicing abstinence or where their partner is sterile (e.g., vasectomy) should be considered to be of childbearing potential.
* Women of child bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of investigational product.
* Female patients within one year of entering the menopause must agree to use an effective non-hormonal method of contraception during the treatment period and for at least 6 months after the last study treatment.
* Males must agree to use an effective method of contraception during the treatment period and for at least 6 months after the last study treatment.
* Absence of any psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up schedule; such conditions should be assessed with the patient before randomization in the trial.
* Before patient randomization and study related procedures (that would not have been performed as part as standard care), written informed consent must be given according to ICH/GCP, and national/local regulations. Informed consent should also be given for biological material to be stored and used for future research on brain tumors.
* Patients with a buffer range from the normal values of +/- 5 % for hematology and +/- 10% for biochemistry are acceptable. A maximum of +/- 2 days for timelines may be acceptable (one day for post operative MRI).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 592 (Actual)
Dates: Start 2011-10 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Time to event

SECONDARY OUTCOMES:
PFS (RANO criteria), median , PFS 6 mo and PFS 12 mo, Overall survival: OS 9,12,24 mo | time to event or fixed time points
Response rate, duration of response and progression pattern | time to event and fixed time points
CTCAE version 4.0. NYHA criteria will be used for assessing heart failure | Worst grade
Patient-oriented criteria: clinical/neurological deterioration free survival, steroid use, quality of life (reported by patients and caregivers/relatives) and development of cognitive deterioration. | 9,12,24 mo
Molecular basis of gliomas and the identification of biomarkers to translate into advances in screening, diagnosis, treatment, and monitoring with improved clinical outcomes | 9,12,24mo

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Wick, Pr., Study Chair — Universitatsklinikum Heidelberg
Locations (2):
- Netherlands (2):
  - Erasmus MC - Daniel den Hoed Cancer Center, Rotterdam
  - Medisch Centrum Haaglanden - Westeinde, The Hague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wick W, Gorlia T, Bendszus M, Taphoorn M, Sahm F, Harting I, Brandes AA, Taal W, Domont J, Idbaih A, Campone M, Clement PM, Stupp R, Fabbro M, Le Rhun E, Dubois F, Weller M, von Deimling A, Golfinopoulos V, Bromberg JC, Platten M, Klein M, van den Bent MJ. Lomustine and Bevacizumab in Progressive Glioblastoma. N Engl J Med. 2017 Nov 16;377(20):1954-1963. doi: 10.1056/NEJMoa1707358. PMID 29141164
- [Derived] Ediebah DE, Reijneveld JC, Taphoorn MJ, Coens C, Zikos E, Aaronson NK, Heimans JJ, Bottomley A, Klein M; EORTC Quality of Life Department and Patient Reported Outcome and Behavioral Evidence (PROBE). Impact of neurocognitive deficits on patient-proxy agreement regarding health-related quality of life in low-grade glioma patients. Qual Life Res. 2017 Apr;26(4):869-880. doi: 10.1007/s11136-016-1426-z. Epub 2016 Oct 15. PMID 27744512